CLINICAL TRIAL: NCT04889716
Title: Phase II Study of Dual Targeting of CD19 and CD20 Antigens Using Sequential CD19-directed CAR-T Cells Followed by Mosunetuzumab or Glofitamab in Relapsed or Refractory Diffuse Large B-cell or Transformed Follicular Lymphomas
Brief Title: CAR-T Followed by Bispecific Antibodies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 48420
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Large B-cell Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — glofitamab; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Cohort 1 subjects will receive mosunetuzumab. Pending demonstrated safety of cohort 1, the trial will progress to cohort 2, in which subjects will receive glofitamab with obinutuzumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Participants receive mosunetuzumab 60 mg for cycles 1 and 2 (although fractionated for cycle 1), and 30 mg for all subsequent cycles after standard-of-care therapy with CD19-directed CAR T-cells
  Interventions: Drug: mosunetuzumab
- Cohort 2 (Experimental): Participants receive obinutuzumab (1000 mg for each subject) and glofitamab after standard-of-care therapy with CD19-directed CAR T-cells. The dose of glofitamab for each subject will be 30 mg, other than for cycle 1, which will be 12.5 mg glofitamab fractionated over two weeks.
  Interventions: Drug: glofitamab; Drug: obinutuzumab

INTERVENTIONS:
Drug: mosunetuzumab — 1 mg IV on Cycle 1 Day 1; 2 mg IV Cycle 1 Day 8; 60 mg IV Cycle 1 Day 15; 60 mg IV on Cycle 2 Day 1 and then 30 mg IV every 21 days beginning Cycle 2 Day 1 through Cycle 17.
  Other Names: RO7030816; BTCT4465A; Lunsumio
  Arms: Cohort 1
Drug: glofitamab — 2.5 mg IV Cycle 1 Day 8; 10 mg IV Cycle 1 Day 15 then 30 mg every 21 days beginning Cycle 2 Day 1 through Cycle 12
  Other Names: CD20 TCB; RO7082859
  Arms: Cohort 2
Drug: obinutuzumab — 1000 mg IV on Cycle 1 Day 1.
  Other Names: Gazyva; Gazyvaro; RO5072759; huMAb <CD20>; GA101
  Arms: Cohort 2

SUMMARY:
The research study is being conducted to test the safety and effectiveness of the experimental drug mosunetuzumab (Cohort 1) or obinutuzumab and glofitamab (Cohort 2) when given after CAR (genetically modified) T cells. The study is for patients who have already received a CAR T-cell infusion. Some patients who join the study will receive mosunetuzumab, other patients later in the study may receive a different experimental drug (glofitamab, in combination with obinutuzumab).

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* History of relapsed or refractory large B-cell lymphoma (including transformed follicular lymphoma, and follicular lymphoma Grade 3B) who have relapsed after or failed to respond to at least one prior standard systemic treatment regimen that contains an anthracycline and at least one containing an anti-CD20-directed therapy and for whom there is no available therapy expected to improve survival (e.g., standard chemotherapy, autologous or allogeneic stem cell transplant).
* PET/CT scan (preferred), diagnostic CT scan, or MRI prior to CAR-T cell therapy, with at least one bi-dimensionally measurable lesion (≥ 1.5 cm for nodal lesion or ≥ 1cm for extra-nodal lesions in largest dimension by low-dose computerized tomography [CT] scan with FDG-uptake ≥ liver); this imaging must have been obtained within 56 days of receiving CAR T cell therapy.
* PET/CT scan (preferred), diagnostic CT scan, or MRI with at least one bi-dimensionally measurable lesion (≥ 1.5 cm for nodal lesion or ≥ 1cm for extra-nodal lesions in largest dimension by low-dose computerized tomography [CT] scan with FDG-uptake ≥ liver); this imaging documenting measurable disease must be obtained at least day +30 after CAR T cell infusion and prior to cycle 1 day 1.
* Be at least 30 days after CAR T-cell infusion at time of study enrollment.
* Adequate laboratory studies,
* Ability and willingness to take proper contraceptive precautions

Exclusion Criteria:

* Had > Grade 3 cytokine release syndrome (CRS) by ASTCT criteria32 after CAR-T therapy or who have unresolved CRS after CAR-T therapy
* Had ≥ grade 2 neurologic toxicity by ASTCT criteria after CAR-T therapy or who have active neurologic toxicity after CAR-T therapy
* Inability to comply with protocol-mandated hospitalization and activities restrictions in the investigators' decision
* Pregnant or lactating, or intending to become pregnant during the study or within 3 months after the last dose of bispecific antibody or 18 months of obinutuzumab, whichever comes later
* Prior solid organ transplantation
* History of autoimmune disease, including but not limited to myocarditis, autoimmune pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, uveitis, vasculitis, or glomerulonephritis
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* History of other malignancy that could affect compliance with the protocol or interpretation of results Significant cardiovascular disease such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina)
* Significant active pulmonary disease (e.g., bronchospasm and/or obstructive pulmonary disease) requiring oxygen or corticosteroid use.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major documented infection requiring treatment with IV antibiotics or hospitalization within 2 weeks prior to first mosunetuzumab or glofitamab administration. Empiric or prophylactic antibiotics administered during neutropenia or neutropenic fever without microbiologic evidence of infection do not exclude patients.
* Recent major surgery within 4 weeks prior to first mosunetuzumab or glofitamab administration
* Active or chronic infection(s) would have increased risks for toxicity if treated with bispecific antibody therapy, thus will be excluded.
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Received systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) with the exception of corticosteroid treatment < 20 mg/day prednisone or equivalent within 2 weeks prior to first dose of bispecific antibody
* History of drug or alcohol abuse within 12 months prior to screening in the investigator's judgment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's and/or Medical Monitor's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the percentage of subjects who achieve a complete metabolic response at 26 weeks from date of first infusion as measured by Cheson 14 (ie Lugano) criteria | 24 weeks from date of first infusion of investigational agent
  Complete response will be assessed using Cheson 2014 or Lugano criteria, utilizing simple 5 point score (Deauville score). For this study complete response will be a score of 1 (no uptake), 2 (uptake ≤ mediastinum), or 3 (uptake >mediastinum but ≤ liver, with no new lesions, and no FDG-uptake in the bone marrow, that is not expected (i.e. due to growth factors or therapy
Assessment of the percentage of subjects who experienced non-hematologic dose limiting toxicity associated with early administration of Mosunetuzumab following SOC CAR-T Cell therapy. | 42 days from the date of first infusion of mosunetuzumab
  DLTs include the following: unexpected ≥grade 3 non-hematologic that is at least possibly related to the study drug, any grade 3 event that does not improve to ≤ grade 2 within 72 hours, any grade 3 AST, ALT or total bilirubin that lasts more than 72 hours in the absence of other causes, ≥ grade 3 neurotoxicity or seizure of any grade.
  Cytokine Relsease Syndrome: CRS grade 4, Grade 3 CRS that does not improve to ≤ grade 2 within 72 hours.
  Grade 1: Temperature ≥ 38°C, no hypotension, no hypoxia. Grade 2: Temperature ≥ 38°C, hypotension not requiring vasopressors and/or hypoxia requiring low flow nasal cannula. Grade 3: Temperature ≥ 38°C, hypotension requiring a vasopressor and/or requiring high flow oxygen. Grade 4: Temperature ≥ 38°C, hypotension requiring multiple vasopressor and/or requiring positive pressure, intubation or mechanical ventilation.
Assessment of the percentage of subjects who experience non-hematologic dose limiting toxicity associated with early administration of glofitimab following SOC CAR-T Cell therapy. | 63 days from the date of first infusion of glofitimab
  Non-hematologic DLTs include the following: unexpected ≥grade 3 non-hematologic that is at least possibly related to the study drug, any grade 3 event that does not improve to ≤ grade 2 within 72 hours, any grade 3 AST, ALT or total bilirubin that lasts more than 72 hours in the absence of other causes, ≥ grade 3 neurotoxicity or seizure of any grade.
  Cytokine Relsease Syndrome: CRS grade 4, Grade 3 CRS that does not improve to ≤ grade 2 within 72 hours.
  Grade 1: Temperature ≥ 38°C, no hypotension, no hypoxia. Grade 2: Temperature ≥ 38°C, hypotension not requiring vasopressors and/or hypoxia requiring low flow nasal cannula. Grade 3: Temperature ≥ 38°C, hypotension requiring a vasopressor and/or requiring high flow oxygen. Grade 4: Temperature ≥ 38°C, hypotension requiring multiple vasopressor and/or requiring positive pressure, intubation or mechanical ventilation.
Assessment of the percentage of subjects who experience hematologic dose limiting toxicity associated with early administration of Mosunetuzumab and glofitimab following SOC CAR-T Cell therapy in patients who stop therapy after 2 cycles. | 63 days from the date of the first infusion or glofitimab or mosunetuzumab
  Dose limiting hematologic toxicities will be measured by the following: ANC < 1000/uL despite G-CSF support, Hgb < 7 g/dL despite transfusion support, Plt < 50,000/uL that lasts for at least 7 days
  Hematologic DLTS that occur within the first 60 days following CAR-T Cell therapy will not be included in this assessment.

SECONDARY OUTCOMES:
Determine Response Duration | from time of first response assessment to up to five years from last dose of bispecific antibody therapy
  Average length of response in months of any partial or complete metabolic responses

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Schuster, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No